CLINICAL TRIAL: NCT03508765
Title: Neurocognitive and Neuroimaging Outcomes in Older Patients With Multiple Myeloma Treated With Autologous Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-154
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: ASCT; Memorial Sloan Kettering Cancer Center; 18-154
MeSH Terms: conditions — Multiple Myeloma | interventions — Magnetic Resonance Imaging; Wechsler Scales; Trail Making Test; Neuropsychological Tests; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- rsfMRI + Neurocognitive Tests (Experimental): Participants diagnosed with multiple myeloma in complete, partial or very good partial remission per standard International Myeloma Working Group Criteria will complete neurocognitive tests and structural and functional rsfMRI (brain MRIs).
  Interventions: Diagnostic Test: Structural Image; Diagnostic Test: Functional Image; Behavioral: Digit Span subtest; Behavioral: Brief Test of Attention; Behavioral: Trail Making Test (Parts A & B); Behavioral: Auditory Consonant Trigrams Test; Behavioral: Controlled Oral Word Association Test; Behavioral: Hopkins Verbal Learning Test-Revised; Behavioral: The Center for Epidemiological Study-Depression; Behavioral: The Functional Assessment of Chronic Illness Therapy-Fatigue Subscale, Version 4; Other: Blood draw

INTERVENTIONS:
Diagnostic Test: Structural Image — Patients will undergo structural and functional (rsfMRI) brain MRIs (total time= ~15 minutes) at enrollment (prior to HD-Chemo/ASCT) and approximately 3-4 months after ASCT.
  Other Names: Brain MRI
Diagnostic Test: Functional Image — Patients will undergo structural and functional (rsfMRI) brain MRIs (total time= ~15 minutes) at enrollment (prior to HD-Chemo/ASCT) and approximately 3-4 months after ASCT.
  Other Names: rsfMRI
Behavioral: Digit Span subtest — Evaluates auditory attention and working memory
  Other Names: WAIS-IV
Behavioral: Brief Test of Attention — Assesses selective auditory attention
  Other Names: BTA
Behavioral: Trail Making Test (Parts A & B) — Assesses visual scanning, graphomotor speed, and setshifting
Behavioral: Auditory Consonant Trigrams Test — Assesses attention and susceptibility to interference
Behavioral: Controlled Oral Word Association Test — A timed test of verbal fluency.
  Other Names: COWAT
Behavioral: Hopkins Verbal Learning Test-Revised — The HVLT-R is a test of verbal learning and recall.
  Other Names: HVLT-R
Behavioral: The Center for Epidemiological Study-Depression — assesses perceived depression
  Other Names: CES-D
Behavioral: The Functional Assessment of Chronic Illness Therapy-Fatigue Subscale, Version 4 — A 13-item questionnaire designed to assess symptoms and concerns specific to the QOL of patients with fatigue
  Other Names: FACIT-FS
Other: Blood draw — Blood samples will be collected at each time point (pre-ASCT; 3-4 months and post-ASCT) to assess serum levels of inflammatory cytokines.

SUMMARY:
The purpose of this study is to learn about possible changes in thinking (cognitive) abilities, such as memory skills, and in brain anatomy and function, in adults with multiple myeloma who are treated with high-dose chemotherapy followed by ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple myeloma and in complete, partial or very good partial remission at enrollment as per standard International Myeloma Working Group Criteria
* Scheduled to have high-dose chemotherapy and ASCT
* Age 60 - 75 years at study entry
* In the judgment of the consenting professional, fluent and able to communicate well enough in English to complete the study assessments and provide informed consent.

  * Patients who report that English is not their primary language will be asked the US Census English proficiency question "How well do you speak English" and the answer "very well" will be required

Exclusion Criteria:

* With signs and/or symptoms of central nervous system cancers (e.g., tumors, metastases, leptomeningial disease) as determined by their physician, medical records, or by a brain MRI, either at the time of enrollment or during the study period
* With current diagnosis of major Axis I psychiatric disorder (DSM-IV), major depression, bipolar disorder, or schizophrenia, as per medical records or patient report
* As per patient report or as confirmed by the medical record, if the patient is taking anti-depression or anti-anxiety medication, < 2 months on these medications or a change in the prescribed dose in the past 2 months
* With history of a neurological disorder, neurodegenerative disease, or traumatic brain injury with loss of consciousness (>60 minutes), as per medical records or patient report
* With a history of another cancer, except for non-melanoma skin cancer, as per medical records or patient report
* With current substance abuse and/or history of substance abuse, as per medical records or patient report
* With evidence of visual or auditory impairment that would preclude completion of the assessments, as per medical records or patient report
* With contraindications to MRI examinations as per standard screening guidelines used in the Department of Radiology (i.e., ferromagnetic material or implants, pacemakers or defibrillators, stents, claustrophobia)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Changes in neurocognitive functions in older participants with Multiple Myeloma following high-dose (HD) chemotherapy and autologous stem cell transplantation (ASCT) assessed by initial and follow-up neurocognitive evaluation | up to 4 months following chemotherapy and ASCT
Changes in regional brain volume and functional connectivity when baseline and follow-up MRIs are compared. | up to 4 months following chemotherapy and ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Denise Correa, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Rutgers University - Data Analysis, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org